CLINICAL TRIAL: NCT03156803
Title: Enhancing Knowledge Translation in Nutrition Through a Healthy Eating Blog: a Randomized Controlled Trial
Brief Title: Enhancing Knowledge Translation in Nutrition Through a Healthy Eating Blog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-257 A3/15-01-2016
Record Dates: First submitted 2016-03-08; First posted 2017-05-17 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy eating blog (HEB) (Experimental): For a 6-month period, mothers randomised to the HEB group will receive a weekly blog post discussing various positive aspects of healthy eating and presenting recipes and strategies to increase dairy product intakes and vegetable and fruit intakes. The posts will be developed with an emphasis of food skills acquisition.
  Interventions: Behavioral: Healthy eating blog
- Control (No Intervention): Mothers randomised to the control group will not have access to the healthy eating blog.

INTERVENTIONS:
Behavioral: Healthy eating blog — For a 6-month period, mothers randomised to the HEB group will receive a weekly blog post discussing various positive aspects of healthy eating and presenting recipes and strategies to increase dairy product intakes and vegetable and fruit intakes. The posts will be developed with an emphasis of food skills acquisition.
  Arms: Healthy eating blog (HEB)

SUMMARY:
The purpose of this study is to evaluate the effects of an evidence-based healthy eating blog on dietary behaviors of mothers

DETAILED DESCRIPTION:
Mothers randomised to the experimental group were exposed to one weekly blog post for 6 months. Blog posts focus on the improvement of dairy products as well as vegetables and fruits consumption targeting five food skills categories: (1) knowledge about food, nutrition and cooking; (2) planning of healthy meals, and for including children to develop their food skills; (3) conceptualizing outcomes; (4) mechanical techniques for food preparation; (5) perception of food characteristics. Each post included a step-by-step recipe developed by the research team and featuring dairy products, vegetables and fruits. Recipes were described textually and also using pictures. Twenty-six posts were created over the six-month intervention. Participants randomised to the control group were not exposed to the healthy eating blog. The primary outcome is the daily intakes of dairy products, vegetables and fruits. The secondary outcomes are mothers' food skills and body weight.

ELIGIBILITY:
Inclusion Criteria:

* Have Internet access, have at least one child aged two to twelve years, are mostly in charge of the planning and preparation of family meals, consume less than two servings a day of dairy products and/or less than seven servings a day of vegetables and fruits.

Exclusion Criteria:

* Take medications that could affect food intake, have eating disorders, are dieting, are currently pregnant or lactating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-10; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Daily intakes of dairy products, vegetables and fruits measured by a validated web-based food frequency questionnaire | 6 months
  Assessed at T=0 month, T=3 months and T=6 months.

SECONDARY OUTCOMES:
Food skills measured by a web-based questionnaire | 6 months
  Food skills measured: planning of healthy meal, knowledge about food, nutrition and cooking, mechanical technics for food preparation, etc. Assessed at T=0 month, T=3 months and T=6 months.
Body weight | 6 months
  Assessed at T=0 month, T=3 months and T=6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Desroches, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dumas AA, Lemieux S, Lapointe A, Provencher V, Robitaille J, Desroches S. Recruitment and retention of mothers of preschoolers and school-aged children in a social media-delivered healthy eating intervention: lessons learned from a randomized controlled trial. Trials. 2020 Aug 10;21(1):706. doi: 10.1186/s13063-020-04628-0. PMID 32778159
- [Derived] Dumas AA, Lemieux S, Lapointe A, Provencher V, Robitaille J, Desroches S. Effects of an Evidence-Informed Healthy Eating Blog on Dietary Intakes and Food-Related Behaviors of Mothers of Preschool- and School-Aged Children: A Randomized Controlled Trial. J Acad Nutr Diet. 2020 Jan;120(1):53-68. doi: 10.1016/j.jand.2019.05.016. Epub 2019 Sep 10. PMID 31519466